CLINICAL TRIAL: NCT05912803
Title: Effects of Simulated Equestrian Therapy on Motor Proficiency and Gait Parameters Among Down Syndrome Children-A Randomized Controlled Trial
Brief Title: Effects of Simulated Equestrian Therapy on Motor Proficiency and Gait Parameters Among Down Syndrome Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Maha Siddiqui, Principal Investigator, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6803223MHREH
Record Dates: First submitted 2023-06-02; First posted 2023-06-22 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulated Equestrian Therapy (Experimental): The treatment group will receive Simulated Equestrian Therapy using 2 horse simulators (wooden and mechanical). Each participant will undergo a warm-up before phase I and cool-down after phase II.
  The treatment will be divided into following 2 phases; Phase I The child will be instructed to ride the mechanical simulator in a pre-defined area measuring 10 yards and complete a total of 4 rounds of this area. Rest periods in between and after will be provided to the child when required. Major muscles of the body will be targeted here to strengthen the core.
  Phase II The child will be instructed to ride the wooden simulator and a combination of goal directed activates will be performed every week for 12 weeks in the following manner;
  0-2 weeks: Practicing catching and throwing.
  3-5 weeks: Placing the ball, and rings on the target.
  6-8 weeks: Target hitting on a game of dart.
  9-12 weeks: Leaning to the head, feet, and tail of the horse
  Interventions: Device: Simulated Equestrian Therapy
- Neuro-Motor Therapy (Active Comparator): This group will perform overall stability and body balancing exercises to strengthen the core and develop the coordination and balance required for task performance. Each activity will be performed in a set of 2-3, considering the activity level of the child, with 8-12 repetitions attaining the available ROM and flexibility of the child thrice for three weeks. The participants will undergo warm-up before the exercise and cool-down afterwards.
  Interventions: Other: Neuro-Motor Therapy

INTERVENTIONS:
Device: Simulated Equestrian Therapy — The treatment group will receive Simulated Equestrian Therapy for 12 weeks thrice per week using 2 horse simulators (wooden and mechanical) in two phases.
  Phase I The child will be instructed to ride the mechanical simulator in a pre-defined area measuring 10 yards and complete a total of 4 rounds of this area. Rest periods in between and after will be provided to the child when required. Major muscles of the body will be targeted here to strengthen the core.
  Phase II The child will be instructed to ride the wooden simulator and a combination of goal directed activates will be performed.
  Arms: Simulated Equestrian Therapy
Other: Neuro-Motor Therapy — This group will perform overall stability and body balancing exercises to strengthen the core and develop the coordination and balance required for task performance. Each activity will be performed in a set of 2-3, considering the activity level of the child, with 8-12 repetitions attaining the available ROM and flexibility of the child. The participants will undergo warm-up before the exercise and cool-down afterwards.
  Arms: Neuro-Motor Therapy

SUMMARY:
According to the World Health Organization (WHO) and United Nations Children's Fund (UNICEF), one billion people suffer from physical and mental disabilities, with 240 million children. Whereas 26.4 million belong to Asia, and approximately 5 million are from Pakistan. The Centre for Disease Control and Prevention (CDC) reports developmental disorders as one of the leading causes of these disabilities. Several conditions are classified under this domain, including Autism Spectrum Disorder, Attention-Deficit Hyperactivity Disorder, Down syndrome, and Cerebral Palsy. Down syndrome (DS) has recently emerged as a prevailing condition in low-and middle-income countries, with an incidence of 1 in every 300 babies. DS is a genetic disorder due to the triplication of all or some parts of the 21st chromosome. Various problems characterize this disability, including; compromised motor skills proficiency and altered gait parameters. These deficits have been addressed using numerous effective techniques, one of which is 'Simulated Equestrian Therapy'. Despite advances in rehabilitating DS patients, a scarcity of literature still surfaces regarding using these simulators and their effects. To our knowledge, no study in Pakistan has been conducted to evaluate motor proficiency and gait parameters in the DS population using this intervention. Therefore, the present study is aimed to assess the effects of simulated equestrian therapy on motor proficiency and gait parameters in DS children.

DETAILED DESCRIPTION:
A total of 58 participants will be recruited for this study after obtaining informed voluntary assent from the guardians. Simple random sampling using the envelop method will be used for the group allocation, to which the participants will be blind. Each participant will be allocated randomly to the treatment group (n=29) that will receive Simulated Equestrian Therapy and the control group (n=29) to receive Neuromotor Therapy. Each participant will be assessed at baseline, after 6 and 12 weeks of intervention using Bruinink's test of motor proficiency (BOT-2) and 10 meter walk test (10MWT). Each participant's blood pressure and heart rate will also be recorded before each session to ensure safety. The participants will be wearing protective gear (belt, helmet, knee and elbow pads) and portable telemetry during the entire session. The session duration in both groups will comprise 30-45 minutes on average, varying with the progression each week. Each session will be provided three times/a week for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with diagnosed DS are referred by a physician.
* Age 6-12 years.
* Ability to independently walk, GMFCS level-I.

Exclusion Criteria:

* Diagnosed atlantoaxial instability.
* Diagnosed osteoarticular, pulmonary or cardiovascular disorders.
* Diagnosed severe behavioral or cognitive impairment.
* Severe visual impairment that cannot be corrected with glasses.
* If equestrian therapy received in the last 1-year.
* Refusal of parents/guardians to participate in the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Bilateral Coordination | Baseline
  Motor proficiency is a combination of 4 skills including; bilateral coordination, balance, speed agility, and strength.
  All of these subsets of motor proficiency are assessed via a battery known as Bruinink's test of motor proficiency, BOT 2. It is a questionnaire that is filled out by the examiner after the successful motor performance of the examinee and scores are given for each attempt. These scores for each subset are summed at the end and a composite score is obtained that indicates the value of motor proficiency of an individual.
Bilateral Coordination | 6 weeks after intervention
  Motor proficiency is a combination of 4 skills including; bilateral coordination, balance, speed agility, and strength.
  All of these subsets of motor proficiency are assessed via a battery known as Bruinink's test of motor proficiency, BOT 2. It is a questionnaire that is filled out by the examiner after the successful motor performance of the examinee and scores are given for each attempt. These scores for each subset are summed at the end and a composite score is obtained that indicates the value of motor proficiency of an individual.
Bilateral Coordination | 12 weeks after intervention
  Motor proficiency is a combination of 4 skills including; bilateral coordination, balance, speed agility, and strength.
  All of these subsets of motor proficiency are assessed via a battery known as Bruinink's test of motor proficiency, BOT 2. It is a questionnaire that is filled out by the examiner after the successful motor performance of the examinee and scores are given for each attempt. These scores for each subset are summed at the end and a composite score is obtained that indicates the value of motor proficiency of an individual.
Balance | Baseline
  Motor proficiency is a combination of 4 skills including; bilateral coordination, balance, speed agility, and strength.
  All of these subsets of motor proficiency are assessed via a battery known as Bruinink's test of motor proficiency, BOT 2. It is a questionnaire that is filled out by the examiner after the successful motor performance of the examinee and scores are given for each attempt. These scores for each subset are summed at the end and a composite score is obtained that indicates the value of motor proficiency of an individual.
Balance | 6 weeks after intervention
  Motor proficiency is a combination of 4 skills including; bilateral coordination, balance, speed agility, and strength.
  All of these subsets of motor proficiency are assessed via a battery known as Bruinink's test of motor proficiency, BOT 2. It is a questionnaire that is filled out by the examiner after the successful motor performance of the examinee and scores are given for each attempt. These scores for each subset are summed at the end and a composite score is obtained that indicates the value of motor proficiency of an individual.
Balance | 12 weeks after intervention
  Motor proficiency is a combination of 4 skills including; bilateral coordination, balance, speed agility, and strength.
  All of these subsets of motor proficiency are assessed via a battery known as Bruinink's test of motor proficiency, BOT 2. It is a questionnaire that is filled out by the examiner after the successful motor performance of the examinee and scores are given for each attempt. These scores for each subset are summed at the end and a composite score is obtained that indicates the value of motor proficiency of an individual.
Speed agility | Baseline
  Motor proficiency is a combination of 4 skills including; bilateral coordination, balance, speed agility, and strength.
  All of these subsets of motor proficiency are assessed via a battery known as Bruinink's test of motor proficiency, BOT 2. It is a questionnaire that is filled out by the examiner after the successful motor performance of the examinee and scores are given for each attempt. These scores for each subset are summed at the end and a composite score is obtained that indicates the value of motor proficiency of an individual.
Speed agility | 6 weeks after intervention
  Motor proficiency is a combination of 4 skills including; bilateral coordination, balance, speed agility, and strength.
  All of these subsets of motor proficiency are assessed via a battery known as Bruinink's test of motor proficiency, BOT 2. It is a questionnaire that is filled out by the examiner after the successful motor performance of the examinee and scores are given for each attempt. These scores for each subset are summed at the end and a composite score is obtained that indicates the value of motor proficiency of an individual.
Speed agility | 12 weeks after intervention
  Motor proficiency is a combination of 4 skills including; bilateral coordination, balance, speed agility, and strength.
  All of these subsets of motor proficiency are assessed via a battery known as Bruinink's test of motor proficiency, BOT 2. It is a questionnaire that is filled out by the examiner after the successful motor performance of the examinee and scores are given for each attempt. These scores for each subset are summed at the end and a composite score is obtained that indicates the value of motor proficiency of an individual.
Strength | Baseline
  Motor proficiency is a combination of 4 skills including; bilateral coordination, balance, speed agility, and strength.
  All of these subsets of motor proficiency are assessed via a battery known as Bruinink's test of motor proficiency, BOT 2. It is a questionnaire that is filled out by the examiner after the successful motor performance of the examinee and scores are given for each attempt. These scores for each subset are summed at the end and a composite score is obtained that indicates the value of motor proficiency of an individual.
Strength | 6 weeks after intervention
  Motor proficiency is a combination of 4 skills including; bilateral coordination, balance, speed agility, and strength.
  All of these subsets of motor proficiency are assessed via a battery known as Bruinink's test of motor proficiency, BOT 2. It is a questionnaire that is filled out by the examiner after the successful motor performance of the examinee and scores are given for each attempt. These scores for each subset are summed at the end and a composite score is obtained that indicates the value of motor proficiency of an individual.
Strength | 12 weeks after intervention
  Motor proficiency is a combination of 4 skills including; bilateral coordination, balance, speed agility, and strength.
  All of these subsets of motor proficiency are assessed via a battery known as Bruinink's test of motor proficiency, BOT 2. It is a questionnaire that is filled out by the examiner after the successful motor performance of the examinee and scores are given for each attempt. These scores for each subset are summed at the end and a composite score is obtained that indicates the value of motor proficiency of an individual.
Cadence | Baseline
  In this study cadence and gait velocity are considered as Parameters of Gait. Both of these parameters are recorded via 10-meter walk test. In this test, the individual walks at their usual comfortable speed at a distance of 10 meters, the speed of walking (gait velocity) is recorded via stopwatch, and the number of steps taken (cadence) are counted as well by the examiner.
Cadence | 6 weeks after intervention
  In this study cadence and gait velocity are considered as Parameters of Gait. Both of these parameters are recorded via 10-meter walk test. In this test, the individual walks at their usual comfortable speed at a distance of 10 meters, the speed of walking (gait velocity) is recorded via stopwatch, and the number of steps taken (cadence) are counted as well by the examiner.
Cadence | 12 weeks after intervention
  In this study cadence and gait velocity are considered as Parameters of Gait. Both of these parameters are recorded via 10-meter walk test. In this test, the individual walks at their usual comfortable speed at a distance of 10 meters, the speed of walking (gait velocity) is recorded via stopwatch, and the number of steps taken (cadence) are counted as well by the examiner.
Gait Velocity | Baseline
  In this study cadence and gait velocity are considered as Parameters of Gait. Both of these parameters are recorded via 10-meter walk test. In this test, the individual walks at their usual comfortable speed at a distance of 10 meters, the speed of walking (gait velocity) is recorded via stopwatch, and the number of steps taken (cadence) are counted as well by the examiner.
Gait Velocity | 6 weeks after intervention
  In this study cadence and gait velocity are considered as Parameters of Gait. Both of these parameters are recorded via 10-meter walk test. In this test, the individual walks at their usual comfortable speed at a distance of 10 meters, the speed of walking (gait velocity) is recorded via stopwatch, and the number of steps taken (cadence) are counted as well by the examiner.
Gait Velocity | 12 weeks after intervention
  In this study cadence and gait velocity are considered as Parameters of Gait. Both of these parameters are recorded via 10-meter walk test. In this test, the individual walks at their usual comfortable speed at a distance of 10 meters, the speed of walking (gait velocity) is recorded via stopwatch, and the number of steps taken (cadence) are counted as well by the examiner.

CONTACTS AND LOCATIONS:
Overall Officials: Sumaira Farooqui, PhD, Study Director — Ziauddin University
Locations (1):
- Ziauddin University and Dar-ul-Sukoon, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No